CLINICAL TRIAL: NCT04343664
Title: Mental Health Assessment Among Community Member During the Covid-19 Pandemic in Indonesia
Acronym: New
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tjhin Wiguna (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor-Investigator, Tjhin Wiguna, Prof. Dr. dr., Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Other Study IDs: MH-Covid19
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Mental Stress; Mental Health Wellness 1; Depression; Anxiety; Behavior Problem; Emotional Problem
Keywords: Mental health, Covid-19, Pandemic, Indonesia
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders; Mental Disorders; Psychological Well-Being; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Covid-19 pandemic in Indonesia makes several changes in daily living. The Indonesian government suggests that everyone should stay at home by implements the work from home and school from home. Therefore, the issues related with Covid-19 are also worrying such as death because of the infection, virus transmission, doing everything from home such as Friday praying for Moslem, Sunday service at home, etc. People is anxious whenever meeting people because they are not really understand whether people is infected or not. Therefore, this study tries to identify the impact of Covid-19 pandemic in Indonesia towards mental well-being of the community.

DETAILED DESCRIPTION:
The Covid-19 pandemic in Indonesia makes several changes in daily living. The Indonesian government suggests that everyone should stay at home by implements the work from home and school from home. Therefore, the issues related with Covid-19 are also worrying such as death because of the infection, virus transmission, doing everything from home such as Friday praying for Moslem, Sunday service at home, etc. People is anxious whenever meeting people because they are not really understand whether people is infected or not. Therefore, this study tries to identify the impact of Covid-19 pandemic in Indonesia towards mental well-being of the community. The aims of this study are trying to collect and identify the most important aspect of mental health that affected by the Covid-19 pandemic in Indonesia, and using this data we are trying to propose the exact mental health promotion and prevention program for the community. The study design is cross sectional. We develop the questionnaire that suitable for our study, consists of demographic data, life experience data. In addition, for assessing mental health problems, the study uses PHQ-9, SRQ-20, GAD-7, SDQ for children 4 - 10 years old and 11 - 17 years old. The study is done by online survey. The data analysis is done by SPSS for mac version 21.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate on this study by signing the informed consent

Exclusion Criteria:

* No

Min Age: 4 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All children, parents and community members
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | up to 5 minutes
  The depression symptoms assessed by Patient Health Queationnaire-9 Scale. The range is 0 -27, the highest score means the highest depresive
Anxiety symptoms | up to 5 minutes
  The anxiety symptoms assessed by Generalized Anxiety Disorder -7 Scale. It is consists of 7 item with ranged score 0 -21. The highest score means the highest anxiety
Stress related problems | up to 7 minutes
  The stress related problems assessed by Self Reporting Questionnaire-20 Scale. The range is 0 -20, the highest score means the highest mental health problems
Behavior and emotional problem among children and adolescents | up to 5 minutes
  Behavior and emotional problem among children and adolescents assessed by Strength and Difficulties Questionnaire. SDQ consists of 25 statements, the score is ranged from 0 - 60. The highest score means the highest problems

CONTACTS AND LOCATIONS:
Overall Officials: Tjhin Wiguna, PhD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital; Tjhin Wiguna, PhD, Principal Investigator — Fakultas Kedokteran Univeristas Indonesia
Locations (1):
- dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Undecided yet